CLINICAL TRIAL: NCT05379504
Title: Reducing COVID-19 Related Disability in Rural Community-Dwelling Older Adults Using Smart Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Rachel Proffitt, Principal Investigator, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2043542; 1R01AG072935-01A1 (NIH)
Record Dates: First submitted 2022-03-21; First posted 2022-05-18 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Quality of Life; Disabilities Multiple
MeSH Terms: interventions — Self-Management

STUDY DESIGN:
Intervention Model Description: Individuals will be randomized to one of two study arms in blocks of 4.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be masked to study participant assignment. Baseline assessments will be completed prior to enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self Management (Experimental): The 5A's Behavior Change Mode [39] is the framework for the self-management intervention. The five "A"s will be addressed through the integration of the self-management intervention and the sensor system. There will be a minimum of four intervention sessions with each healthcare profession (OT, RN, and SW) for 12 visits per participant.
  Interventions: Behavioral: Self Management
- Health Education (Active Comparator): Participant's randomized to the standard health education arm will receive the intervention at Month 1 and then months 3, 6, 9 and 12.
  Interventions: Behavioral: Standard Health Education

INTERVENTIONS:
Behavioral: Standard Health Education — Participants randomized to the standard health education arm will receive the intervention at month 1 and then months 3, 6, 9, and 12 (coinciding with the quarterly interviews). The participant will use the tablet and telehealth platform to complete the interview and education session with research staff. The content of these sessions will be focused on helping the participant (and family member/caregiver as appropriate) understand their health data, assisting them with any technology issues and providing the participant with education on their condition(s) and any requested resources. Research staff will will also provide any additional health education if there are changes to conditions or new diagnoses after an outside provider visit.
  Arms: Health Education
Behavioral: Self Management — The self-management intervention will be delivered over the course of a year. There will be a minimum of four intervention sessions with each healthcare profession (OT, RN and SW) for 12 visits per participant. The team (OT, RN and SW) will meet twice during the first 2 months to determine a lead interventionist based on the participant's SMART goals and areas of concern. The lead interventionist will have three additional sessions with the participant and will be the point-person for sensor system alerts and messages. Goal Attainment Scaling [83] will be administered during the quarterly interview to assess participant progress on SMART goals. This measure is administered collectively with the participant, provides further accountability, offers opportunities to the participant for reflection on progress, and is a concrete measure of "success" of the self-management intervention.
  Arms: Self Management

SUMMARY:
The social distancing requirements for COVID-19 coupled with the adverse health impacts of social isolation and decreased access to healthcare in rural areas places older adults with disabilities in a dire situation. The smart sensor system to be deployed and studied in this project aims to reduce disability for rural community-dwelling older adults and improve health-related quality of life, including depression and anxiety. An implementation guide will be developed to increase success of future scale-up evaluations.

DETAILED DESCRIPTION:
Over 85% of Missouri is rural and individuals in these rural areas are older and have reduced access to regular healthcare as compared to individuals living in urban areas of Missouri. Those with disabilities, particularly older adults, are at higher risk for contracting COVID-19. There is a critical need to reduce disability and improve quality of life for community-dwelling older adults with disabilities for successful aging-in-place during the COVID-19 pandemic. The investigators have developed, with our partner company Foresite Healthcare, a proven sensor-based technology solution for monitoring health-related behaviors in the home. In a multi-site randomized controlled trial, the investigators demonstrated that the sensor system with nursing care coordination prevents declines in function for older adults living in assisted living facilities. The long-term goal of this research is to support independent living for older adults with disabilities for as long as possible. The purpose of this project is to deploy the sensor system in the homes of rural community-dwelling older adults with disabilities and evaluate the effect of the sensor system on reducing disability and improving health-related quality of life. Using a two-arm randomized controlled trial, the sensor system will be installed in the homes of 64 older adults. Participants randomized to Study Arm 1 will receive a multidisciplinary (nursing, occupational therapy, and social work) self-management intervention paired with the sensor system. This intervention is based on the 5As self-management approach and is a direct translation of the nursing care coordination in our prior research. Participants randomized to Study Arm 2 will have standard health education paired with the sensor system. An implementation guide for future use with different partner agencies will be developed using individual and setting level data collected from Aims 1, 2 and 3 using the RE-AIM framework. The project will be accomplished in three aims. In Aim 1, the investigators will evaluate the effect of a sensor system paired with a multidisciplinary self-management intervention as compared to the sensor system paired with standard health education care on disability and health-related quality of life after 1 year. In Aim 2, the investigators will evaluate the effect of the sensor system on secondary health outcomes (depression, anxiety, occupational performance, and caregiver burden), rates of falls, and healthcare usage. In Aim 3, the investigators will collect individual participant data for satisfaction and adoption and stakeholder data about organizational setting. Data from Aims 1, 2 and 3 will be analyzed using RE-AIM to produce implementation guidance contextualized by organizational setting. For older adults with disabilities living in rural areas, the sensor system has the potential to change the approach to healthcare and disability management.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 65, Live in a rural defined county, Have difficulty with at least 1 self-care task or 2 daily living tasks, Have internet access, Able to stand with or without assistance

Exclusion Criteria:

* Life expectancy less than one year, Severe cognitive impairment (mini mental state exam score <17), Life in a facility that provides care services, Katz ADL Score of 6, Receiving in-home physical therapy, occupational therapy or nursing, Have been hospitalized more than three times in teh previous 12 months, Plan to change residences within the next year

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Katz ADL Index | 1 year
  Disability
Change in PROMIS-29 | 1 year
  Health-related quality of life

SECONDARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale | 1 year
  Depression and anxiety
Change in Canadian Occupational Performance Measure | 1 year
  Occupational performance
Change in Patient Activation Measure | 1 year
  Patient activation/self-efficacy
Technology Experience Profile | Baseline
  Experience with technology

CONTACTS AND LOCATIONS:
Overall Officials: Rachel M Proffitt, OTD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share de-identified clinical outcome data and parameters extracted from the sensor system (e.gs., motion density, gait speed) associated with the study participants by depositing these data at the National Archive of Computerized Data on Aging (NACDA) which is an NIH-funded repository. Submitted data will confirm with relevant data and terminology standards. Data will be de-identified following the University of Missouri IRB procedures. All sensor parameters are stored on the secure server as de-identified data so no further processing will be required before depositing at NACDA. Identifiers will be removed from clinical outcome data before depositing at NACDA. All personal and private information of study participants will be protected using our secure data collection system (RedCap) on an encrypted network. No personal or private information will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available at the completion of the study and will be held according to parameters for the National Archive of Computerized Data on Aging (NACDA)
Access Criteria: As I will be using National Archive of Computerized Data on Aging (NACDA), which is an NIH-funded repository, this repository has policies and procedures in place that will provide data access to qualified researchers, fully consistent with NIH data sharing policies and applicable laws and regulations.
URL: http://www.icpsr.umich.edu/web/pages/NACDA/index.html

REFERENCES:
- [Background] Missouri Department of Health and Senior Services 2019. Health in rural Missouri: Biennial report 2018-2019. http://health.mo.gov/living/families/ruralhealth/pdf/biennial2019.pdf
- [Background] Research and Training Center on Disability in Rural Communities. 2020. Missouri State Profile. http://rtc.ruralinstitute.umt.edu/state-profile-map-series/missouri-state-profile/
- [Background] Kane, R, L, (1999). A new model of chronic care. Generations-Journal of the American Society on Aging, 23(2), 35-37
- [Background] Rantz M, Phillips LJ, Galambos C, Lane K, Alexander GL, Despins L, Koopman RJ, Skubic M, Hicks L, Miller S, Craver A, Harris BH, Deroche CB. Randomized Trial of Intelligent Sensor System for Early Illness Alerts in Senior Housing. J Am Med Dir Assoc. 2017 Oct 1;18(10):860-870. doi: 10.1016/j.jamda.2017.05.012. Epub 2017 Jul 12. PMID 28711423
- [Background] Rantz MJ, Scott SD, Miller SJ, Skubic M, Phillips L, Alexander G, Koopman RJ, Musterman K, Back J. Evaluation of health alerts from an early illness warning system in independent living. Comput Inform Nurs. 2013 Jun;31(6):274-80. doi: 10.1097/NXN.0b013e318296298f. PMID 23774449
- [Background] Rantz MJ, Skubic M, Miller SJ, Galambos C, Alexander G, Keller J, Popescu M. Sensor technology to support Aging in Place. J Am Med Dir Assoc. 2013 Jun;14(6):386-91. doi: 10.1016/j.jamda.2013.02.018. Epub 2013 Apr 3. PMID 23562281
- [Background] Skubic M, Guevara RD, Rantz M. Automated Health Alerts Using In-Home Sensor Data for Embedded Health Assessment. IEEE J Transl Eng Health Med. 2015 Apr 10;3:2700111. doi: 10.1109/JTEHM.2015.2421499. eCollection 2015. PMID 27170900
- [Background] Skubic, M., Guevara, R. D., & Rantz, M. (2012). Testing classifiers for embedded health assessment. Proc., International Conference on Smart Homes and Health Telematics, Artimino, Italy, pp. 198-205
- [Background] Jain, A., Keller, J., & Popescu, M. (2019, June 23-26). Explainable Al for dataset comparison, {Paper presentation}. 2019 IEEE International Conference on Fuzzy Systems (FUZZ-IEEE).
- [Background] Ibrahim, O. A., Keller, J., & Popescu, M. (2019) An unsupervised framework for detecting early signs of illness in eldercare. [Paper presentation}. 2019 IEEE International Conference on Bioinformatics and Biomedicine (BIBM), San Diego, CA, USA
- [Background] Ibrahim, O.A., Keller, J.M., & Popescu, M. (2017). Context preserving representation of daily activities in elder care. {Paper presentation}. IEEE International Conference on Bioinformatics and Biomedicine (BIBM)
- [Background] Ibrahim, O.A., Popescu, M., & Keller, J.M. (2017). Unsupervised Analysis of Activity Patterns in Eldercare Monitoring. {Paper presentation}. American Medical Informatics Association (AMIA) Annual Symposium.
- [Background] Wu, W., Keller, J.M., Skubic, M., Popescu, M., & Lane, K.R. (in review). Early detection of health changes in the elderly using in-home multi-sensors data streams.
- [Background] Mishra, A.K., Skubic, M., Despins, L.A., Popescu, M., Rantz, M., Keller, J., & Lane, K. (2019). Development of a functional health index for older adults using the electronic health record. {Paper presentation}. IEEE EMBS International Conference on Biomedical & Health Informatics (BHI), Chicago, IL, United States.
- [Background] Robinson EL, Park G, Lane K, Skubic M, Rantz M. Technology for Healthy Independent Living: Creating a Tailored In-Home Sensor System for Older Adults and Family Caregivers. J Gerontol Nurs. 2020 Jul 1;46(7):35-40. doi: 10.3928/00989134-20200605-06. PMID 32597999
- [Background] Shelani, S., Levins, T., Robinson, E.L., Lane, K., Park, G., & Skubic, M. (2019). Development and comparison of customized voice-assistant systems for independent living older adults {Paper presentation}. HCII conference, Orlando, FL, United States
- [Background] Federal Interagency Forum on Aging Related Statistics. (2016). Older Americans 2016: Key Indicators of Wellbeing. Washington DC: US Government Printing Office.
- [Background] He, W., Larsen, L. J., and U.S. Census Bureau. (2014, December). Older Americans with a disability. Washington, DC, U.S. Government Printing Office.
- [Background] Griffith L, Raina P, Wu H, Zhu B, Stathokostas L. Population attributable risk for functional disability associated with chronic conditions in Canadian older adults. Age Ageing. 2010 Nov;39(6):738-45. doi: 10.1093/ageing/afq105. Epub 2010 Sep 1. PMID 20810673
- [Background] Fong JH. Disability incidence and functional decline among older adults with major chronic diseases. BMC Geriatr. 2019 Nov 21;19(1):323. doi: 10.1186/s12877-019-1348-z. PMID 31752701
- [Background] Center for Disease Control and Prevention. (2012). Preventing Chronic disease. Multiple Chronic Conditions Among US Adults; A2012 Update. Retrieved from http://www.cdc.gov/pcd/issues/2014/13_0389.htm Accessed May 15, 2020.
- [Background] U.S. Administration on Aging. (2014). A Profile of Older Americans; 2014. Department of Health and Human Services Washington, DC, Retrieved from http://www.aoa.acl.gov/Aging_Statistics/Profile/2014/docs/2014-Profile.pdf. Accessed May 15, 2020.
- [Background] Herbert C, Molinsky JH. What Can Be Done To Better Support Older Adults To Age Successfully In Their Homes And Communities? Health Aff (Millwood). 2019 May;38(5):860-864. doi: 10.1377/hlthaff.2019.00203. Epub 2019 Apr 24. PMID 31017475
- [Background] Santos-Eggimann B, Meylan L. Older Citizens' Opinions on Long-Term Care Options: A Vignette Survey. J Am Med Dir Assoc. 2017 Apr 1;18(4):326-334. doi: 10.1016/j.jamda.2016.10.010. Epub 2016 Dec 9. PMID 27956072
- [Background] Skinner HG, Coffey R, Jones J, Heslin KC, Moy E. The effects of multiple chronic conditions on hospitalization costs and utilization for ambulatory care sensitive conditions in the United States: a nationally representative cross-sectional study. BMC Health Serv Res. 2016 Mar 1;16:77. doi: 10.1186/s12913-016-1304-y. PMID 26926525
- [Background] Schoen C, Davis K, Willink A. Medicare Beneficiaries' High Out-of-Pocket Costs: Cost Burdens by Income and Health Status. Issue Brief (Commonw Fund). 2017 May;11:1-14. PMID 28498650
- [Background] Banerjee D. The impact of Covid-19 pandemic on elderly mental health. Int J Geriatr Psychiatry. 2020 Dec;35(12):1466-1467. doi: 10.1002/gps.5320. Epub 2020 Jun 27. No abstract available. PMID 32364283
- [Background] Armitage R, Nellums LB. COVID-19 and the consequences of isolating the elderly. Lancet Public Health. 2020 May;5(5):e256. doi: 10.1016/S2468-2667(20)30061-X. Epub 2020 Mar 20. No abstract available. PMID 32199471
- [Background] Steinman MA, Perry L, Perissinotto CM. Meeting the Care Needs of Older Adults Isolated at Home During the COVID-19 Pandemic. JAMA Intern Med. 2020 Jun 1;180(6):819-820. doi: 10.1001/jamainternmed.2020.1661. No abstract available. PMID 32297903
- [Background] Beutel ME, Klein EM, Brahler E, Reiner I, Junger C, Michal M, Wiltink J, Wild PS, Munzel T, Lackner KJ, Tibubos AN. Loneliness in the general population: prevalence, determinants and relations to mental health. BMC Psychiatry. 2017 Mar 20;17(1):97. doi: 10.1186/s12888-017-1262-x. PMID 28320380
- [Background] Boyle CA, Fox MH, Havercamp SM, Zubler J. The public health response to the COVID-19 pandemic for people with disabilities. Disabil Health J. 2020 Jul;13(3):100943. doi: 10.1016/j.dhjo.2020.100943. Epub 2020 May 24. PMID 32499132
- [Background] Turk MA, McDermott S. The COVID-19 pandemic and people with disability. Disabil Health J. 2020 Jul;13(3):100944. doi: 10.1016/j.dhjo.2020.100944. Epub 2020 May 28. No abstract available. PMID 32475803
- [Background] Rantz M, Skubic M, Abbott C, Galambos C, Popescu M, Keller J, Stone E, Back J, Miller SJ, Petroski GF. Automated In-Home Fall Risk Assessment and Detection Sensor System for Elders. Gerontologist. 2015 Jun;55 Suppl 1(Suppl 1):S78-87. doi: 10.1093/geront/gnv044. PMID 26055784
- [Background] Rantz M, Lane K, Phillips LJ, Despins LA, Galambos C, Alexander GL, Koopman RJ, Hicks L, Skubic M, Miller SJ. Enhanced registered nurse care coordination with sensor technology: Impact on length of stay and cost in aging in place housing. Nurs Outlook. 2015 Nov-Dec;63(6):650-5. doi: 10.1016/j.outlook.2015.08.004. Epub 2015 Sep 8. PMID 26463735
- [Background] Galambos C, Rantz M, Back J, Jun JS, Skubic M, Miller SJ. Older Adults' Perceptions of and Preferences for a Fall Risk Assessment System: Exploring Stages of Acceptance Model. Comput Inform Nurs. 2017 Jul;35(7):331-337. doi: 10.1097/CIN.0000000000000330. PMID 28187009
- [Background] Connelly K, Molchan H, Bidanta R, Siddh S, Lowens B, Caine K, Demiris G, Siek K, Reeder B. Evaluation framework for selecting wearable activity monitors for research. Mhealth. 2021 Jan 20;7:6. doi: 10.21037/mhealth-19-253. eCollection 2021. PMID 33634189
- [Background] Glasgow RE, Funnell MM, Bonomi AE, Davis C, Beckham V, Wagner EH. Self-management aspects of the improving chronic illness care breakthrough series: implementation with diabetes and heart failure teams. Ann Behav Med. 2002 Spring;24(2):80-7. doi: 10.1207/S15324796ABM2402_04. PMID 12054323
- [Background] Wagner EH, Davis C, Schaefer J, Von Korff M, Austin B. A survey of leading chronic disease management programs: are they consistent with the literature? Manag Care Q. 1999 Summer;7(3):56-66. PMID 10620960
- [Background] Glasgow RE, Orleans CT, Wagner EH. Does the chronic care model serve also as a template for improving prevention? Milbank Q. 2001;79(4):579-612, iv-v. doi: 10.1111/1468-0009.00222. PMID 11789118
- [Background] Rantz M, Popejoy LL, Galambos C, Phillips LJ, Lane KR, Marek KD, Hicks L, Musterman K, Back J, Miller SJ, Ge B. The continued success of registered nurse care coordination in a state evaluation of aging in place in senior housing. Nurs Outlook. 2014 Jul-Aug;62(4):237-46. doi: 10.1016/j.outlook.2014.02.005. Epub 2014 Feb 22. PMID 24731918
- [Background] Boockvar KS, Lachs MS. Predictive value of nonspecific symptoms for acute illness in nursing home residents. J Am Geriatr Soc. 2003 Aug;51(8):1111-5. doi: 10.1046/j.1532-5415.2003.51360.x. PMID 12890074
- [Background] Boockvar K, Brodie HD, Lachs M. Nursing assistants detect behavior changes in nursing home residents that precede acute illness: development and validation of an illness warning instrument. J Am Geriatr Soc. 2000 Sep;48(9):1086-91. doi: 10.1111/j.1532-5415.2000.tb04784.x. PMID 10983908
- [Background] Hogan J. Why don't nurses monitor the respiratory rates of patients? Br J Nurs. 2006 May 11-24;15(9):489-92. doi: 10.12968/bjon.2006.15.9.21087. PMID 16723921
- [Background] Ridley S. The recognition and early management of critical illness. Ann R Coll Surg Engl. 2005 Sep;87(5):315-22. doi: 10.1308/003588405X60669. PMID 16176687
- [Background] Mann DM, Chen J, Chunara R, Testa PA, Nov O. COVID-19 transforms health care through telemedicine: Evidence from the field. J Am Med Inform Assoc. 2020 Jul 1;27(7):1132-1135. doi: 10.1093/jamia/ocaa072. PMID 32324855
- [Background] Laver KE, Schoene D, Crotty M, George S, Lannin NA, Sherrington C. Telerehabilitation services for stroke. Cochrane Database Syst Rev. 2013 Dec 16;2013(12):CD010255. doi: 10.1002/14651858.CD010255.pub2. PMID 24338496
- [Background] Varnfield M, Karunanithi M, Lee CK, Honeyman E, Arnold D, Ding H, Smith C, Walters DL. Smartphone-based home care model improved use of cardiac rehabilitation in postmyocardial infarction patients: results from a randomised controlled trial. Heart. 2014 Nov;100(22):1770-9. doi: 10.1136/heartjnl-2014-305783. Epub 2014 Jun 27. PMID 24973083
- [Background] Piotrowicz E, Baranowski R, Bilinska M, Stepnowska M, Piotrowska M, Wojcik A, Korewicki J, Chojnowska L, Malek LA, Klopotowski M, Piotrowski W, Piotrowicz R. A new model of home-based telemonitored cardiac rehabilitation in patients with heart failure: effectiveness, quality of life, and adherence. Eur J Heart Fail. 2010 Feb;12(2):164-71. doi: 10.1093/eurjhf/hfp181. Epub 2009 Dec 30. PMID 20042423
- [Background] Little, L., Wallisch, A., Pope, E., & Dunn, W. (2018). Acceptability and cost comparison of telehealth intervention for families of children with autism.
- [Background] Little, L., Wallisch, A., Pope, El, & Dunn, W. (2018). Acceptability and cost comparison of a telehealth intervention for families of children with autism. Infants and Young Children. 31(4), 275-286
- [Background] Weisz, J.R. (2015). Bridging the research-practice divide in youth psychotherapy. The deployment-focused model and transdiagnostic treatment. Verhaltenstherapie, 25(2), 129-132
- [Background] Wainer, A.L., Dvortcsak, A., & Ingersoll, B. (2018). Designing for Dissemination: The Utility of the Deployment. Handbook of Parent-implemented interventions for a Very Young Children with Autism, 425
- [Background] Wang, S. (2011). Change Detection for Eldercare Using Passive Sensing. PhD. Thesis, Electrical and Computer Engineering Dept., University of Missouri, Columbia, MO
- [Background] Wang S, Skubic M, Zhu Y. Activity density map visualization and dissimilarity comparison for eldercare monitoring. IEEE Trans Inf Technol Biomed. 2012 Jul;16(4):607-14. doi: 10.1109/TITB.2012.2196439. Epub 2012 Apr 25. PMID 22547460
- [Background] Wang S, Skubic M, Zhu Y, Galambos C. Using Passive Sensing to Estimate Relative Energy Expenditure for Eldercare Monitoring. Proc IEEE Int Conf Pervasive Comput Commun. 2011 Mar 21:642-648. doi: 10.1109/PERCOMW.2011.5766968. PMID 25266777
- [Background] Heise D, Skubic M. Monitoring pulse and respiration with a non-invasive hydraulic bed sensor. Annu Int Conf IEEE Eng Med Biol Soc. 2010;2010:2119-23. doi: 10.1109/IEMBS.2010.5627219. PMID 21096574
- [Background] Heise D, Rosales L, Skubic M, Devaney MJ. Refinement and evaluation of a hydraulic bed sensor. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:4356-60. doi: 10.1109/IEMBS.2011.6091081. PMID 22255304
- [Background] Rosales, L., Bo-Yu, S., Skkubic, M. & Ho, K.C. (2017). Heart rate estimation from hydraulic bed sensor ballistocardiogram. Journal of Ambient Intelligence and Smart Environments, 9(2), 193-207
- [Background] Lydon K, Su BY, Rosales L, Enayati M, Ho KC, Rantz M, Skubic M. Robust heartbeat detection from in-home ballistocardiogram signals of older adults using a bed sensor. Annu Int Conf IEEE Eng Med Biol Soc. 2015;2015:7175-9. doi: 10.1109/EMBC.2015.7320047. PMID 26737947
- [Background] Starr, I., Rawson, A., Schroeder, H., & Joseph, N. (1939). Studies on the estimation of cardiac output in man, and of abnormalities in cardiac function , from the heart's recoil and the blood's impacts; the ballistocardiogram, American Journal of Physiology--Legacy Content, 127 (1), 1-28
- [Background] Stone, E., & Skubic, M. (2011). Evaluation of an inexpensive depth camera for in-home gait assessment. Journal of Ambient Intelligence and Smart Environments, 3(4), 349-361.
- [Background] Stone EE, Skubic M. Unobtrusive, continuous, in-home gait measurement using the Microsoft Kinect. IEEE Trans Biomed Eng. 2013 Oct;60(10):2925-32. doi: 10.1109/TBME.2013.2266341. Epub 2013 Jun 5. PMID 23744661
- [Background] Stone EE, Skubic M, Back J. Automated health alerts from Kinect-based in-home gait measurements. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:2961-4. doi: 10.1109/EMBC.2014.6944244. PMID 25570612
- [Background] Banerjee T, Keller JM, Skubic M. Resident identification using kinect depth image data and fuzzy clustering techniques. Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:5102-5. doi: 10.1109/EMBC.2012.6347141. PMID 23367076
- [Background] Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the Timed Up & Go Test. Phys Ther. 2000 Sep;80(9):896-903. PMID 10960937
- [Background] Stone E, Skubic M, Rantz M, Abbott C, Miller S. Average in-home gait speed: investigation of a new metric for mobility and fall risk assessment of elders. Gait Posture. 2015 Jan;41(1):57-62. doi: 10.1016/j.gaitpost.2014.08.019. Epub 2014 Sep 6. PMID 25245308
- [Background] Stone EE, Skubic M. Fall detection in homes of older adults using the Microsoft Kinect. IEEE J Biomed Health Inform. 2015 Jan;19(1):290-301. doi: 10.1109/JBHI.2014.2312180. Epub 2014 Mar 17. PMID 24733032
- [Background] Phillips LJ, DeRoche CB, Rantz M, Alexander GL, Skubic M, Despins L, Abbott C, Harris BH, Galambos C, Koopman RJ. Using Embedded Sensors in Independent Living to Predict Gait Changes and Falls. West J Nurs Res. 2017 Jan;39(1):78-94. doi: 10.1177/0193945916662027. Epub 2016 Jul 28. PMID 27470677
- [Background] Proffitt R, Glegg S, Levac D, Lange B. End-user involvement in rehabilitation virtual reality implementation research. J Enabling Technol. 2019;13(2):92-100. doi: 10.1108/JET-10-2018-0050. Epub 2019 Jun 17. PMID 31663039
- [Background] Proffitt R, Lange B, Chen C, Winstein C. A comparison of older adults' subjective experiences with virtual and real environments during dynamic balance activities. J Aging Phys Act. 2015 Jan;23(1):24-33. doi: 10.1123/japa.2013-0126. Epub 2013 Dec 11. PMID 24334299
- [Background] Proffitt R, Lange B. Feasibility of a Customized, In-Home, Game-Based Stroke Exercise Program Using the Microsoft Kinect(R) Sensor. Int J Telerehabil. 2015 Nov 20;7(2):23-34. doi: 10.5195/ijt.2015.6177. eCollection 2015 Fall. PMID 27563384
- [Background] Reeder B, Chung J. Joe J, Lazar A, Thompson HJ, Demiris G. Understanding Older Adults' Perceptions of IN-Home Sensors Using an Obtrusiveness Framework. HCI International 2016; July 17-22, 2016; Toronto CA: Springer; 2016
- [Background] Reeder B, Chung J, Le T, Thompson H, Demiris G. Assessing older adults' perceptions of sensor data and designing visual displays for ambient environments. An exploratory study. Methods Inf Med. 2014;53(3):152-9. doi: 10.3414/ME13-02-0009. Epub 2014 Apr 14. PMID 24728081
- [Background] Reeder B, Chung J, Lazar A, Joe J, Demiris G, Thompson HJ. Testing a theory-based mobility monitoring protocol using in-home sensors: a feasibility study. Res Gerontol Nurs. 2013 Oct;6(4):253-63. doi: 10.3928/19404921-20130729-02. Epub 2013 Aug 5. PMID 23938159
- [Background] Pak, R, & McLaughlin, A. (2010). Designing displays for older adults: CRC Press
- [Background] Fisk AD, Rogers WA, Charness N, Czaja SJ, & Sharit J. (2009). Designing for older adults: Principles and creative human factors approaches. Boca Raton, FL: CRC press
- [Background] Shelkey M, Wallace M. Katz Index of Independence in Activities of Daily Living (ADL). Director. 2000 Spring;8(2):72-3. No abstract available. PMID 11081028
- [Background] Suijker JJ, Buurman BM, ter Riet G, van Rijn M, de Haan RJ, de Rooij SE, Moll van Charante EP. Comprehensive geriatric assessment, multifactorial interventions and nurse-led care coordination to prevent functional decline in community-dwelling older persons: protocol of a cluster randomized trial. BMC Health Serv Res. 2012 Apr 1;12:85. doi: 10.1186/1472-6963-12-85. PMID 22462516
- [Background] Szanton, S.L., & Gitlin, L.N. (2016). Meeting the health care financing imperative through focusing on function. The CAPABLE studies. Public Policy & Aging Report. 26(3), 106-110
- [Background] Hays RD, Spritzer KL, Schalet BD, Cella D. PROMIS(R)-29 v2.0 profile physical and mental health summary scores. Qual Life Res. 2018 Jul;27(7):1885-1891. doi: 10.1007/s11136-018-1842-3. Epub 2018 Mar 22. PMID 29569016
- [Background] Deyo RA, Katrina Ramsey, Buckley DI, Michaels L, Kobus A, Eckstrom E, Forro V, Morris C. Performance of a Patient Reported Outcomes Measurement Information System (PROMIS) Short Form in Older Adults with Chronic Musculoskeletal Pain. Pain Med. 2016 Feb;17(2):314-24. doi: 10.1093/pm/pnv046. PMID 26814279
- [Background] Lewis, T.F., Larson, M.F., & Korcuska, J.S. (2017). Strengthening the planning process of motivational interviewing using goal attainment scaling. Journal of Mental Health Counseling, 39(3), 195-210
- [Background] Gearing RE, El-Bassel N, Ghesquiere A, Baldwin S, Gillies J, Ngeow E. Major ingredients of fidelity: a review and scientific guide to improving quality of intervention research implementation. Clin Psychol Rev. 2011 Feb;31(1):79-88. doi: 10.1016/j.cpr.2010.09.007. Epub 2010 Oct 7. PMID 21130938
- [Background] Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003 Aug 1;1:29. doi: 10.1186/1477-7525-1-29. PMID 12914662
- [Background] Cup EH, Scholte op Reimer WJ, Thijssen MC, van Kuyk-Minis MA. Reliability and validity of the Canadian Occupational Performance Measure in stroke patients. Clin Rehabil. 2003 Jul;17(4):402-9. doi: 10.1191/0269215503cr635oa. PMID 12785249
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Background] Barg-Walkow, L.H., Mitzner, T.L., & ROgers, W.A. (2014). Technology Experience Profile (TEP): Assessment and Scoring Guide. HFA-TR-1402). Atlanta, GA: Georgia Institute of Technology, School of Psychology, Human Factors and Aging Laboratory.
- [Background] Green LW, Glasgow RE, Atkins D, Stange K. Making evidence from research more relevant, useful, and actionable in policy, program planning, and practice slips "twixt cup and lip". Am J Prev Med. 2009 Dec;37(6 Suppl 1):S187-91. doi: 10.1016/j.amepre.2009.08.017. No abstract available. PMID 19896017
- [Background] Glasgow RE, Klesges LM, Dzewaltowski DA, Bull SS, Estabrooks P. The future of health behavior change research: what is needed to improve translation of research into health promotion practice? Ann Behav Med. 2004 Feb;27(1):3-12. doi: 10.1207/s15324796abm2701_2. PMID 14979858
- [Background] Boyatzis RE. Thematic analysis and code development: Transforming qualitative information. London and New Delhi: Sage Publications. 1998
- [Background] Turner AM, Reeder B, Ramey J. Scenarios, personas and user stories: user-centered evidence-based design representations of communicable disease investigations. J Biomed Inform. 2013 Aug;46(4):575-84. doi: 10.1016/j.jbi.2013.04.006. Epub 2013 Apr 22. PMID 23618996
- [Background] Reeder B, Turner AM. Scenario-based design: a method for connecting information system design with public health operations and emergency management. J Biomed Inform. 2011 Dec;44(6):978-88. doi: 10.1016/j.jbi.2011.07.004. Epub 2011 Jul 23. PMID 21807120
- [Background] Reeder B, Zaslavksy O, Wilamowska KM, Demiris G, Thompson HJ. Modeling the oldest old: personas to design technology-based solutions for older adults. AMIA Annu Symp Proc. 2011;2011:1166-75. Epub 2011 Oct 22. PMID 22195177
- [Background] Reeder B, Hills RA, Turner AM, Demiris G. Participatory design of an integrated information system design to support public health nurses and nurse managers. Public Health Nurs. 2014 Mar-Apr;31(2):183-92. doi: 10.1111/phn.12081. Epub 2013 Sep 30. PMID 24117760
- [Background] Reeder B, Demiris G. Building the PHARAOH framework using scenario-based design: a set of pandemic decision-making scenarios for continuity of operations in a large municipal public health agency. J Med Syst. 2010 Aug;34(4):735-9. doi: 10.1007/s10916-009-9288-3. Epub 2009 Apr 23. PMID 20703929